CLINICAL TRIAL: NCT05227339
Title: RAE (Realize, Analyze, Engage)- A Digital Biomarker Based Detection and Intervention System for Stress and Craving During Recovery From Substance Use Disorder: Phase II
Brief Title: RAE (Realize, Analyze, Engage)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ContinueYou, LLC (Industry)
Collaborators: University of Massachusetts, Worcester (Other); University of Texas at Tyler (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RAEPHASEII
Record Dates: First submitted 2022-01-25; First posted 2022-02-07 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Substance Use Disorders; Treatment Adherence and Compliance
Keywords: mhealth; stress; craving; wearables; technology; digital diagnostics; digital health
MeSH Terms: conditions — Substance-Related Disorders; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Interventional (RAE + Usual Care) (Experimental): Subjects will receive usual care through an outpatient substance use disorder treatment facility, will be provided with a wearable sensor and the RAE mobile application. Participants will be instructed to use the RAE app for a minimum of 30 days.
  Interventions: Device: RAE
- Control (Usual care) (No Intervention): Subjects will receive usual care through an outpatient substance use disorder treatment facility and will be provided with a wearable sensor (fitness tracker). They will not be given access to the RAE mobile app.

INTERVENTIONS:
Device: RAE — Subjects in the interventional group will have access to the RAE Health mobile app which receives continuous physiologic data from a wearable device. Algorithms embedded in the RAE app detect stress and craving events, and trigger mobile phone notifications when detected. Notifications are paired to real-time mindfulness based interventions.
  Other Names: RAE Mobile App
  Arms: Interventional (RAE + Usual Care)

SUMMARY:
The proposed study will evaluate the detection of digital biomarkers of stress, and drug craving in a population of individuals undergoing treatment for substance use disorder

DETAILED DESCRIPTION:
RAE integrates digital detection of high-risk stress and craving periods by utilizing a mobile phone application and integrated wearable sensor. These detections are paired with interventions (mindfulness based de-escalation tools), support, and monitoring (to identify trends and plan for future). The present study will deploy the technology in a multi-site randomized controlled trial to test the efficacy of the RAE system in on clinical and psychosocial outcomes. Subjects will be randomized to use the RAE system (mobile app and wearable sensor) plus usual care vs usual care plus a fitness tracker only to measure differences retention in treatment, return to substance use, and overall psychosocial functioning. The ultimate goal is to develop a cost-effective, paradigm changing recovery tool that will improve substance use disorder treatment, and prevent related complications and deaths.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Enrolled in an outpatient SUD treatment program
* Enrolled in treatment for < 90 days
* Fluent in English
* Have access to a smartphone with iOS or Android Capabilities
* Capable of providing informed consent

Exclusion Criteria:

* Pregnancy
* Prisoner Status
* Significant limitation of range of motion of non-dominant arm (amputation or fracture)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with return to drug use | 3 months
  Relapse to use of substance use defined as 1) self-reported use, 2) positive urine drug screen (from treatment program) or 3) provider report of confirmed relapse (Only applies to substances for which subject is receiving treatment)

SECONDARY OUTCOMES:
Number of participants retained in treatment | 3 months
  Participants status as engaged in recovery treatment (index treatment program or other)
Number of hospitalizations and emergency department visits per participant | 3 months
  Includes absolute number of Emergency Department visits (SUD and non-SUD related), number of unplanned hospital admissions (SUD and non-SUD related), number of days hospitalized (SUD and non-SUD related admissions) and overdose related visits

CONTACTS AND LOCATIONS:
Overall Officials: Megan Reinhardt, Principal Investigator — ContinueYou, LLC
Locations (1):
- University of Massachusetts Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carreiro S, Taylor M, Shrestha S, Reinhardt M, Gilbertson N, Indic P. Realize, Analyze, Engage (RAE): A Digital Tool to Support Recovery from Substance Use Disorder. J Psychiatr Brain Sci. 2021;6:e210002. doi: 10.20900/jpbs.20210002. Epub 2021 Feb 24. PMID 33748430
- [Background] Carreiro S, Chintha KK, Shrestha S, Chapman B, Smelson D, Indic P. Wearable sensor-based detection of stress and craving in patients during treatment for substance use disorder: A mixed methods pilot study. Drug Alcohol Depend. 2020 Apr 1;209:107929. doi: 10.1016/j.drugalcdep.2020.107929. Epub 2020 Mar 3. PMID 32193048